CLINICAL TRIAL: NCT07154927
Title: Evaluation of the Feasibility of Ultrasonography Guided Pulmonary Artery Catheterization in Pulmonary Hypertension Diagnosis.Pulmonary Artery Catheters (PACs) That Called Swan-Ganz Catheters Provide Valuable Information in Select Patient's Especially Pulmonary Hypertension Patiens. PACs Are Indicated for Assessment of Cardiopulmonary Hemodynamics in Specific Groups of Patients Presenting With Pulmonary Hypertension, Pulmonary Embolism or Shock [1]. They Can be Inserted at Bedside Under Sterile Conditions and Provide Valuable Information That Can Add Benefit for Measures Recorded With Transthor
Brief Title: Evaluation of Feasibility of Ultrasonography Guided Pulmonary Artery Catheterization in Pulmonary Hypertension Diagnosis
Status: Not yet recruiting | Type: Observational
Sponsor: Mostafa K. Ahmed (Other)
Responsible Party: Sponsor-Investigator, Mostafa K. Ahmed, Assiut University Faculty of Medicine chest departement pulmonary hypertension Unit, Assiut University
Organization: Assiut University (Other)
Other Study IDs: ASSIUTMOSTAFAKAHMED
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary artery catheterization , ultrasonography guidance
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pulmonary artery catheters (PACs) that called Swan-Ganz catheters provide valuable information in select patient's especially pulmonary hypertension patiens. PACs are indicated for assessment of cardiopulmonary hemodynamics in specific groups of patients presenting with pulmonary hypertension, pulmonary embolism or shock [1]. They can be inserted at bedside under sterile conditions and provide valuable information that can add benefit for measures recorded with transthoracic echocardiography. The advancement of PACs in a patient is usually performed by flotation of a balloon tipped catheter under pressure waveform guidance. The balloon tip floats in blood and is directed into the pulmonary artery by the normal flow from superior vena cava and through the right heart chambers into pulmonary artery. The correct positioning is needed for safe use and accurate cardiopulmonary hemodynamics measurement. The use of blind approach of insertion can be challenging in patients with slow blood flow as pulmonary hypertension patients. The abnormal flow can induce the PAC to coil in cardiac chambers such as right atrium and right ventricle or be misdirected to the inferior vena cava. Repeated attempts to retract and redirect the catheter can increase the risk of complications and should be avoided [2]. The use of fluoroscopic guidance persists in these cases. Fluoroscopy when used alongside pressure waveform analysis has been noted to reduce the time to wedge, number of attempts and composite complication rate in patients undergoing pulmonary hemodynamic assessment. Also, fluoroscopy provides real time visualization that can lead to reduction of catheter malposition and ventricular arrhythmias. Unfortunately, it is not available in all pulmonary hypertension units for bedside insertion and hemodynamics evaluation. The use of fluoroscopy can led to unnecessary radiation exposure to both the patient and the procedure team. Sonographic guided pulmonary catheter insertion is interesting technique ; however it still needed to be studied in pulmonary hypertension patients in pulmonary hypertension unit

DETAILED DESCRIPTION:
pulmonary artery catheterization for hemodynamics assessment patients with suggestion of having certain pulmonary hypertensions groups is vital for establishing their managements; few tools are used to facilitate catheter insertion including monitor waves form, fluoroscopic guidance and to lesser extent sonographics guidance. sonographic guidance is not fully studied in pulmonary hypertenison patients however it carries advantages over radiographic guidance of being less exposure to radiation for both the patients and health care team. with increasing pulmonary hypertension units allover the worlds and patients recognitions in addition to availability of ultrasonography that necessitate this study to evaluate sonographic guidance in pulmonary hypertension patients

ELIGIBILITY:
Inclusion Cr### **Inclusion Criteria**

* Adults (≥18 years)
* Clinically suspected PH referred for diagnostic RHC
* Informed consent provided

  ### **Exclusion Criteria**
* Hemodynamic instability requiring immediate intervention
* Poor echocardiographic window despite TTE/TEE
* Contraindications to catheterization
* Known intracardiac shunts or severe tricuspid regurgitation (if it impairs catheter tracking)

iteria: -

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pulmonary hypertension patients refered to our pulmonary hyperetnsion unit for PAC
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Success rate** of PAC placement using ultrasound guidance alone | procedure time from starting patient puncture till procedure end (PAC)
  Time to catheter placement (in minutes)
  * Incidence of complications (major and minor)
  * Accuracy of hemodynamic parameters compared to standard reference
  * Learning curve evaluation over time

CONTACTS AND LOCATIONS:
Overall Officials: mostafa K Ahmed, MD, Principal Investigator — Assiut University pulmonary hypertension Unit Chest Department

IPD SHARING:
Plan to Share IPD: Undecided